CLINICAL TRIAL: NCT01748331
Title: The Significance of the Vasopressin System of the Hemodynamics, Water Balance and Prognosis in Chronic Heart Failure
Brief Title: The Effect of Fluid Restriction in Congestive Heart Failure Complicated With Hyponatremia
Acronym: Decongest
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Finn Gustafsson (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Finn Gustafsson, Staff Cardiologist, PhD, DMSci, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-1-2012-060
Record Dates: First submitted 2012-12-10; First posted 2012-12-12 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure; Hyponatremia
Keywords: Heart Failure; Hyponatremia; Fluid restriction
MeSH Terms: conditions — Heart Failure; Hyponatremia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strict fluid restriction < 1 L/day (Other): 20 patients will be randomized to strict fluid restriction < 1 L/day
  Interventions: Other: Fluid restriction
- Moderate fluid restriction < 2.5 L/day (Other): 20 patients will be randomized to moderate fluid restriction < 2.5 L/day
  Interventions: Other: Fluid restriction

INTERVENTIONS:
Other: Fluid restriction — Patients will be randomized to strict fluid restriction < 1 L/day versus moderate fluid restriction < 2.5 L/day

SUMMARY:
The purpose of this study is to determine the effect of fluid restriction and the neurohormonal mechanisms in the development of hyponatremia in patients with congestive heart failure and hyponatremia. The hypothesis is that strict fluid restriction leads to a larger increase in plasma sodium than standard treatment in patients with decompensated heart failure associated with hyponatremia. A secondary hypothesis is that the neurohormonal change is greater in patients treated with strict fluid restriction versus standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Left Ventricular Ejection Fraction (LVEF) < 40

At least two of the following signs of decompensated heart failure and fluid retention:

* Weight gain > 2 kg
* Pulmonal Congestion
* Jugular vein congestion
* Peripheral oedemas
* Hepatic congestion with ascites
* Radiographic signs of fluid retention
* Increased diuretic dose

And

* New York Heart Association (NYHA) class III-IV
* Plasma sodium < 135 mmol/L
* Symptomatic heart failure and treatment with relevant heart failure medications (beta-blocker, diuretic, digoxin, angiotensin-converting-enzyme inhibitor, angiotensin-II receptor antagonist, spironolactone, hydralazine and/or nitrates)for at least 1 month
* Hospitalization for decompensated heart failure within the last 48 hours
* Given informed consent

Exclusion Criteria:

* Plasma sodium ≥ 135 mmol/L before randomization
* Reduced kidney function (creatinine > 200 μmol/L)
* Severe hematologic disease
* Hypovolemic hyponatremia (volume depletion or dehydration)
* Intolerability to large or fast changes in fluid volume assessed by the investigator
* Plasma sodium < 120 mmol/L accompanied by neurologic symptoms
* Anuria
* Symptomatic systolic blood pressure (supine systolic blood pressure < 90 mmHg)
* Uncontrolled hypertension (systolic blood pressure > 180 mmHg)
* Uncontrolled diabetes diabetes mellitus
* Adrenal insufficiency
* Acute myocardial infarction, sustained ventricular tachycardia or ventricular fibrillation within the last 30 days
* Heart surgery within the last 60 days
* Other severe heart disease: hypertrophic cardiomyopathy, severe heart valve disease, cardiac amyloidosis, active myocarditis, pericardial exudate which is hemodynamically significant
* Left ventricular assist device (LVAD)
* Planned revascularization procedure, electrophysiologic device implantation, mechanic left ventricular assist device, heart transplant or any other heart surgery procedures within the next 30 days
* Cerebrovascular event within the last 6 months
* Comorbidity with an expected survival < 6 months
* Other reasons for hyponatremia: Primary syndrome of inappropriate antidiuretic hormone secretion (SIADH), primary polydipsia, head trauma, uncontrolled hypothyroidism, adrenal insufficiency or other known pharmacologically triggered hyponatremia which is reversible upon discontinuation of the drug, hyperglycemia (pseudohyponatremia), present abuse of alcohol
* Pregnancy
* Pregnant or fertile women who are not using safe contraception
* Dementia
* Unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Change in plasma sodium from day 1 to day 4: - Normalization of plasma sodium or - A significant change in plasma sodium of a minimum of 5 mmol/L from baseline to day 4 | 5 days

SECONDARY OUTCOMES:
Change in plasma vasopressin and copeptin | 5 days
Change in blood pressure, heart rate, weight and oedemas | 5 days
Change in dyspnoea assessed by the patient | 5 days
Number of days until clinical stability | 5 days
The correlation between hospitalization time and plasma sodium | 5 days
Correlation between fluid restriction and change in kidney function | 5 days
Patient assessment of fluid restriction | 5 days
Patient compliance to fluid restriction | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Finn Gustafsson, MD, PhD, DMSci, Principal Investigator — Department of Cardiology, Copenhagen University Hospital, Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Department of Cardiology, Copenhagen University Hospital, Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen